CLINICAL TRIAL: NCT00109213
Title: Greenwich Lumbar Stenosis SLIP Study: A Multi-center, Randomized, Prospective Clinical Trial Comparing Spinal Laminectomy to Laminectomy With Instrumented Pedicle Screw Fusion for Lumbar Stenosis With Grade I Spondylolisthesis
Brief Title: Greenwich Lumbar Stenosis SLIP Study
Acronym: SLIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Greenwich Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GH-SLIP-384
Record Dates: First submitted 2005-04-26; First posted 2005-04-26 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Spinal Stenosis; Spondylolisthesis
Keywords: Spinal Stenosis; Lumbar Spine; Decompression; Fusion; Spondylolisthesis; Prospective, randomized clinical trial
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Lumbar Laminectomy without Fusion
  Interventions: Procedure: Lumbar Laminectomy
- 2 (Active Comparator): Lumbar Laminectomy with Pedicle Screw Instrumented Fusion
  Interventions: Procedure: Lumbar Laminectomy with Instrumented Pedicle Screw Fusion

INTERVENTIONS:
Procedure: Lumbar Laminectomy with Instrumented Pedicle Screw Fusion — Removal of bone to decompress spinal nerves with placement of spinal screws and extra bone to strengthen the spine
  Arms: 2
Procedure: Lumbar Laminectomy — Removal of bone to decompress spinal nerves
  Arms: 1

SUMMARY:
The purpose of the study is to determine the proper use of lower back screws and rods (instrumentation) and bony fusion in subjects with one level of degenerative spinal narrowing (stenosis) compressing nerves to the legs with one spinal bone slipping forward on another (spondylolisthesis). There are two types of operations that surgeons perform for this problem. Some spinal surgeons remove some bone in the back (laminectomy) to decompress the nerves. Other surgeons perform a laminectomy (decompression) as above, but feel that it is also important to strengthen the back by placing screws and rods into the spine and adding more bone to obtain a new bridge of bone away from the nerves (decompression with instrumented fusion). This study aims to test the hypothesis that adding instrumented fusion to a decompression for this spinal problem will improve long term patient outcomes.

DETAILED DESCRIPTION:
There is considerable debate among spinal surgeons regarding the optimal surgical procedure for lumbar spinal stenosis with a grade I spondylolisthesis. The major question is whether or not instrumented pedicle screw fusion should be undertaken when a decompressive laminectomy is performed to relieve neural compression. This multi-center, randomized, prospective clinical study aims to address this question by testing the hypothesis that adding instrumented fusion to a decompression for this spinal problem will improve long-term patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic lumbar spinal stenosis and single level grade I spondylolisthesis (3-14 mm)

Exclusion Criteria:

* History of previous lumbar spinal surgery in region of stenosis
* Gross spinal instability (defined as greater than 3 mm motion on flexion/extension studies)
* Serious medical illness (ASA Class III or higher)
* Spondylolisthesis greater than 14 mm or associated with spondylolysis

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2002-05; Primary Completion 2009-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
SF-36 (physical component summary score) | 2 year

SECONDARY OUTCOMES:
Oswestry Disability Index | 2 year, 3 year, 4 year
Major Complication rate | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Ghogawala, MD, Study Director — Yale University School of Medicine (Greenwich Hospital); Edward C Benzel, MD, Study Director — Cleveland Clinic Spine Institute (Cleveland Clinic Foundation)
Locations (5):
- United States (5):
  - Greenwich Hospital, Greenwich, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Cleveland Clinic Spine Institute, Cleveland, Ohio
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Background] Ghogawala Z, Benzel EC, Amin-Hanjani S, Barker FG 2nd, Harrington JF, Magge SN, Strugar J, Coumans JV, Borges LF. Prospective outcomes evaluation after decompression with or without instrumented fusion for lumbar stenosis and degenerative Grade I spondylolisthesis. J Neurosurg Spine. 2004 Oct;1(3):267-72. doi: 10.3171/spi.2004.1.3.0267. PMID 15478364
- [Background] Fischgrund JS, Mackay M, Herkowitz HN, Brower R, Montgomery DM, Kurz LT. 1997 Volvo Award winner in clinical studies. Degenerative lumbar spondylolisthesis with spinal stenosis: a prospective, randomized study comparing decompressive laminectomy and arthrodesis with and without spinal instrumentation. Spine (Phila Pa 1976). 1997 Dec 15;22(24):2807-12. doi: 10.1097/00007632-199712150-00003. PMID 9431616
- [Background] Herkowitz HN, Kurz LT. Degenerative lumbar spondylolisthesis with spinal stenosis. A prospective study comparing decompression with decompression and intertransverse process arthrodesis. J Bone Joint Surg Am. 1991 Jul;73(6):802-8. PMID 2071615
- [Derived] Ghogawala Z, Dziura J, Butler WE, Dai F, Terrin N, Magge SN, Coumans JV, Harrington JF, Amin-Hanjani S, Schwartz JS, Sonntag VK, Barker FG 2nd, Benzel EC. Laminectomy plus Fusion versus Laminectomy Alone for Lumbar Spondylolisthesis. N Engl J Med. 2016 Apr 14;374(15):1424-34. doi: 10.1056/NEJMoa1508788. PMID 27074067
- [Derived] Ghogawala Z, Schwartz JS, Benzel EC, Magge SN, Coumans JV, Harrington JF, Gelbs JC, Whitmore RG, Butler WE, Barker FG 2nd. Increased Patient Enrollment to a Randomized Surgical Trial Through Equipoise Polling of an Expert Surgeon Panel. Ann Surg. 2016 Jul;264(1):81-6. doi: 10.1097/SLA.0000000000001483. PMID 26501698
- [Derived] Blumenthal C, Curran J, Benzel EC, Potter R, Magge SN, Harrington JF Jr, Coumans JV, Ghogawala Z. Radiographic predictors of delayed instability following decompression without fusion for degenerative grade I lumbar spondylolisthesis. J Neurosurg Spine. 2013 Apr;18(4):340-6. doi: 10.3171/2013.1.SPINE12537. Epub 2013 Feb 1. PMID 23373567